CLINICAL TRIAL: NCT00089167
Title: Risk Adapted Intravenous Melphalan and Adjuvant Thalidomide and Dexamethasone for Untreated Patients With Primary Systemic Amyloidosis
Brief Title: Melphalan, Thalidomide, and Dexamethasone in Treating Patients With Newly Diagnosed, Previously Untreated Primary Systemic Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 02-031; MSKCC-02031
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: primary systemic amyloidosis
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Immunoglobulin Light-chain Amyloidosis | interventions — Filgrastim; Dexamethasone; Melphalan; Thalidomide

INTERVENTIONS:
Biological: filgrastim
Drug: dexamethasone
Drug: melphalan
Drug: thalidomide

SUMMARY:
RATIONALE: Drugs such as melphalan, thalidomide, and dexamethasone may be effective in treating patients with primary systemic amyloidosis.

PURPOSE: This phase II trial is studying how well giving melphalan together with thalidomide and dexamethasone works in treating patients with primary systemic amyloidosis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 2-year and overall progression-free survival of patients with newly diagnosed, previously untreated primary systemic (AL) amyloidosis treated with risk-adapted melphalan followed by thalidomide and dexamethasone.

Secondary

* Determine plasma cell disease response in these patients at 3, 12, and 24 months after treatment with this regimen.
* Determine amyloid-related disease response in these patients at 12 and 24 months after treatment with this regimen.
* Determine the prognostic significance of immunoglobulin light-chain variable-region germline gene expression by AL plasma cell clones in patients treated with this regimen.
* Determine whether there is molecular minimal residual disease at 12 and 24 months in patients achieving a complete hematologic response after treatment with this regimen.

OUTLINE: Patients are stratified according to the extent of amyloid-related disease (low-risk vs high-risk).

* High-risk disease: Patients receive 2 courses of low-dose melphalan IV, dexamethasone, and filgrastim (G-CSF). After 3 months, patients receive thalidomide and dexamethasone if plasma cell disease persists.
* Low-risk disease: Patients receive 1 course of high-dose melphalan IV and G-CSF. Patients then receive thalidomide and dexamethasone as in high-risk disease regimen.

Patients are followed at 3, 12, and 24 months.

PROJECTED ACCRUAL: A total of 82 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of primary systemic (AL) amyloidosis within the past 12 months

  * High- or low-risk disease, determined by the extent of systemic organ involvement with disease and patient age

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* SWOG 0-3

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* No New York Heart Association class III or IV congestive heart failure
* No restrictive cardiomyopathy requiring oxygen
* No myocardial infarction within the past 6 months
* No symptomatic cardiac arrhythmia within the past 60 days

Other

* No other active malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I cancer in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for AL amyloidosis

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No other prior or concurrent therapy for AL amyloidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-05; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Overall progression-free survival at 2 years

SECONDARY OUTCOMES:
Plasma cell disease response at 3, 12, and 24 months after treatment
Amyloid-related disease response at 12 and 24 months after treatment
Prognostic significance of immunoglobulin light-chain variable-region germline gene expression by AL cell clones
Molecular minimal residual disease at 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Raymond L. Comenzo, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Madhav Dhodapkar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Cohen AD, Zhou P, Reich L, et al.: Risk-adapted intravenous melphalan followed by adjuvant dexamethasone (D) and thalidomide (T) for newly diagnosed patients with Systemic AL Amyloidosis (AL): interim results of a phase II study. [Abstract] Blood 104 (11): A-542, 2004.